CLINICAL TRIAL: NCT05807646
Title: Effect of Ligation Sequence of the Inferior Mesenteric Artery and Vein on Circulating Tumor Cells and Survival in Laparoscopic Rectal Cancer Surgery: a Prospective, Multicenter, Randomized Controlled Study (ARVECTS)
Brief Title: Reduced Dissemination of Tumor Cells With Primary Ligation of the Inferior Mesenteric Vein in Rectal Cancer Patients.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Collaborators: Sichuan Provincial People's Hospital (Other); The Second People's Hospital of Chengdu (Other)
Responsible Party: Principal Investigator, Tao Pan, Principal Investigator, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SichuanCHRI123
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vein ligation first (Experimental): During this procedure, patients undergo laparoscopic rectal cancer surgery with the inferior mesenteric vein ligated first.
  Interventions: Other: Vein ligation first
- Artery ligation first (Active Comparator): During this procedure, patients undergo laparoscopic rectal cancer surgery with the inferior mesenteric artery ligated first.
  Interventions: Other: Artery ligation first

INTERVENTIONS:
Other: Vein ligation first — During this procedure, patients undergo laparoscopic rectal cancer surgery with the inferior mesenteric vein ligated first.
  Arms: Vein ligation first
Other: Artery ligation first — During this procedure, patients undergo laparoscopic rectal cancer surgery with the inferior mesenteric artery ligated first.
  Arms: Artery ligation first

SUMMARY:
Effect of ligation sequence of the inferior mesenteric artery and vein on circulating tumor cells and survival in laparoscopic rectal cancer surgery: a prospective, multicenter, randomized controlled study (ARVECTS)

DETAILED DESCRIPTION:
Several studies have demonstrated that the presence of circulating tumor cells (CTCs) in the peripheral blood can be a surrogate biomarker to predict recurrence and prognosis of rectal cancer. CTCs are released from the primary tumor into the bloodstream and have the potential to spread to distant sites and develop into micro-metastatic deposits. Numerous studies have demonstrated that surgical manipulation could promote the dissemination of tumor cells into the circulation. Theoretically, the potential risk of tumor cell dissemination can theoretically be minimized if the effluent vein was ligated first. However, there is no regulation in the current guidelines on the sequence of ligation of the inferior mesenteric artery and vein during rectal cancer surgery owing to a lack of sufficient evidence. This multi-center randomized controlled trial is to investigate effect of ligation sequence of the inferior mesenteric artery and vein on circulating tumor cells and survival in laparoscopic rectal cancer surgery

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years;
2. Histopathologically confirmed as rectal adenocarcinoma(tumor located within 15 cm from the anal verge at colonoscopy);
3. Patients with a stage I-III rectal cancer eligible for surgery and R0 resection is expected, patients with pelvic lateral lymph nodes metastasis are ineligible;
4. ECOG score: 0-1;
5. ASA score: I/II/III;
6. Laparoscopic surgery;
7. Informed consent.

Exclusion Criteria:

1. Patients who have received preoperative treatment (such as preoperative radiotherapy and chemotherapy);
2. Receiving transanal total mesorectal excision (taTME), specimen extraction through natural lumen (NOSES) ;
3. Recurrent rectal cancer;
4. Simultaneous or metachronous colorectal cancer;
5. Malignant tumors of other organs in the past 5 years or at the same time;
6. The results of preoperative physical examination and imaging examination showed that: (1) the tumor involved the surrounding organs and required combined organ resection; (2) distant metastasis; (3) could not be resected at R0;
7. Pregnant or lactating women;
8. Patients with severe mental disorder;
9. It is not suitable for patients undergoing laparoscopic surgery (such as extensive adhesion caused by previous abdominal surgery or inability to tolerate artificial pneumoperitoneum);
10. History of unstable angina pectoris or myocardial infarction in the past 6 months;
11. Have a history of cerebrovascular accident in the past 6 months;
12. Systemic administration of corticosteroids within 1 month before enrollment;
13. Taking folic acid related drugs within half a year before operation.
14. Severe cardiac insufficiency (FEV1<50% of predicted values);
15. Emergency surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The changes of the level of circulating tumor cells in the peripheral blood | During the surgery
  The changes of the level of circulating tumor cells in the peripheral blood before cutting the skin and after closing the abdomen

SECONDARY OUTCOMES:
3-year disease-free survival | From date of surgery, assessed up to 36 months
  The proportion of patients with no disease recurrence and metastasis after 3 years of surgery
3-years overall survival | From date of surgery, assessed up to 36 months
  The proportion of patients who survived 3 years after surgery
Recurrence pattern | From date of surgery, assessed up to 36 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type
Blood loss | During the surgery
  Blood loss during the surgery
Operation time | During the surgery
  Operation time
Conversive rate | During the surgery
  Conversive rate
Number of lymph nodes collected | During the surgery
  Number of lymph nodes collected
Intraoperative morbidity and mortality rates | During the surgery
  The intraoperative morbidity rates are defined as the rates of event observed within operation
Postoperative morbidity and motality rates | 30 days
  This is for the early postoperative complication, which defined as the event observed within 30 days after surgery
Postoperative recovery course | 10 days
  Time to first ambulation, flatus, liquid diet and soft diet, duration of postoperative hospital stay and postoperative pain are used to assess the postoperative recovery course.Visual analog pain score method is used to evaluate the difference of postoperative pain degree

CONTACTS AND LOCATIONS:
Overall Officials: Chao Liu, Professor, Study Director — Sichuan Cancer Hospital and Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan T, Hu H, Liu C, Zhou HY. Effect of ligation sequence of the inferior mesenteric artery and vein on circulating tumour cells and survival in minimally invasive rectal cancer surgery: study protocol for a randomised controlled trial (ARVECTS study). BMJ Open. 2025 Nov 19;15(11):e098428. doi: 10.1136/bmjopen-2024-098428. PMID 41263842